CLINICAL TRIAL: NCT00695097
Title: The Effect of Rituximab on the Development of Anti-Donor Antibodies and Resolution of B Cell Infiltration in the Renal Allograft of Patients Undergoing Rejection
Brief Title: The Effect of Rituximab on the Development of Anti-Donor Antibodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GNE Rituxin
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Renal Transplant Rejection
Keywords: Rituximab; Renal Transplant Rejection; B cells; Patients with biopsy proven acute rejection cellular infiltrate, B cells
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Rituximab Group: The Rituximab dose is 1000mg (1gm) given as an IV infusion every two weeks for 2 doses (days 1 and 15) and followed up monthly for 1 year. Biopsy was done Baseline and Month 3 and other labs (CBC/Diff, Platelets, HACA, PK, Serum Creatinine, 24-hour protein, HLA antibodies, flow cytometry, and serology testing). Physical exam and vital signs were done.
  Interventions: Drug: Rituximab
- 2 (Active Comparator): No Rituximab: received standard immunosuppression and was followed up monthly for 1 year. Labs (CBC/Diff, Platelets, HACA, PK, Serum Creatinine, 24-hour protein, HLA antibodies, flow cytometry, and serology testing) vital signs, and physical exam was done.
  Interventions: Drug: No Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab infusion on Day 1 and Day 15
  Other Names: Rituxan
  Arms: 1
Drug: No Rituximab — No Rituximab
  Arms: 2

SUMMARY:
The aim of the study is to find out if Rituximab, which is an antibody against specific white cells involved in rejection, when combined with standard anti-rejection treatment can more effectively reverse the rejection process.

Our hypothesis is that with acute rejection there is activation of B cells and the subsequent development of anti-donor antibodies that ultimately lead to graft loss. More effective therapy targeted at B cells may abort the development of anti-HLA antibodies, prevent renal injury and have a favorable effect on long-term graft outcome.

DETAILED DESCRIPTION:
This is a two center, randomized pilot study of the effects of Rituximab on treatment of acute rejection. A total of 24 patients (including patients transplanted at University of California San Francisco and University of Alabama Birmingham) will be enrolled in the study, 16 randomized to Rituximab and 8 to no-Rituximab (control arm). Fifteen (15) subjects will be recruited at UCSF with 10 patients randomized to Rituximab and 5 to no-Rituximab (control arm). If either center is a slow enroller the patient mix could be altered.

Procedures:

This is an open label trial of patients with rejection with B cell infiltrates on kidney biopsy who will be randomized to either receive Rituximab or no Rituximab in and 2:1 ratio. Patients who have rejection on kidney biopsy and on immunohistochemistry there is evidence of B cells infiltration will be enrolled in the study and randomized 2:1 to receive Rituximab or no Rituximab. Rituximab will be administered in 2 doses of 1,000 mg. The first dose will be administered while the patient is still in the hospital being treated for rejection and the second dose will be administered 2 weeks later in the outpatient facility in the GCRC at UCSF. The patients' acute rejection episode will be treated according to standard therapy as per the treating transplant physician. Below is the table (table 1) detailing when the patient will have blood drawn for flow cytometry, anti-HLA antibodies, PK studies, serum creatinine as well as 24 hour urine protein. At 3 months after enrollment in the study, the patient will undergo a follow-up biopsy to determine the extent of the resolution of the cellular infiltrate.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a kidney transplant or kidney-pancreas transplant with predominant findings on kidney biopsy of acute rejection and the presence of as B cells by immunohistochemistry
* Patients between 18 and 65 years of age
* Patients known not to be allergic to Rituximab
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Adequate renal function as indicated by serum creatinine less than 6 mg/dL
* negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.
* Patients who have received a kidney-pancreas transplant.
* Patients who on immunohistochemistry have evidence of B cell infiltration

Exclusion Criteria:

* Patients who have undergoing multi-organ transplant except for kidney-pancreas patients.
* Patients who have been administered an experimental drug in the 3 months preceding enrollment in the study
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera® / Rituxan®)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of HIV (positive HIV, HIV conducted during screening if applicable)
* History of Hepatitis B and/or Hepatitis C (Hep B/C at screening)
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment)
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma insitu of the cervix.
* History of psychiatric disorder being treated with medications
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease) Laboratory Exclusion Criteria (at Screening)
* Hemoglobin: < 7 gm/dL
* Platelets: < 100,000/mm
* Known history of positive Hepatitis B or C serology
* Known history of positive HIV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF-Kidney Transplant Clinic, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients with biopsy-proven ACR were recruited in the kidney transplant Clinic at UCSF and were randomized to either the Rituximab or the control group.
Pre-assignment Details: 18 patients were consented to participate. 3 patients failed eligibility screening prior to treatment assignment. 15 were eligible, 10 were in the Rituximab group and 5 in the no-Rituximab group.
Groups:
- Rituximab Group: Rituximab Group: Rituximab dose is 1000 mg given as an IV infusion every 2 weeks (day 1 and 15) and followed monthly for 1 year.
- Control Group: No Rituximab; Standard maintenance immunosuppressive regimen only and being followed monthly for 1 year.
Period: Overall Study
Arm/Group | Rituximab Group | Control Group
Started | 10 | 5
Completed | 9 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol
Groups:
- Rituximab Group: Rituximab Group: The Rituximab dose is 1000mg (1gm) given as an IV infusion every two weeks for 2 doses (days 1 and 15) and followed monthly for 1 year.
- Control Group: No Rituximab; Standard maintenance immunosuppressive regimen only followed up monthly for 1 year.
- Total: Total of all reporting groups
Arm/Group | Rituximab Group | Control Group | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Biopsy Cell Densities From Baseline to Follow-up
Description: Follow-up biopsy was done 3-6 months after study treatment. Study follow-up monthly for 1 year.
Time Frame: 1 year
Population: 5 Rituximab participants and 4 Control participants provided both baseline and follow-up biopsies for analysis. 6 participants withdrew their consent.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- Rituximab Group: Rituximab infusion day 1 and 15
- Control Group: No Rituximab infusion
Arm/Group | Rituximab Group | Control Group
Number analyzed (Participants) | 5 | 4
cells/mm^3
  CD3 | -164 (0.25) | -122.5 (0.46)
  CD20 | -129.4 (0.054) | 30.4 (0.062)
Statistical Analysis 1: Comparison: Rituximab Group; Pretreatment (Baseline)compared to post-treatment (follow-up) CD3 cell density; Test type: Superiority or Other; p = 0.25, t-test, 2 sided — P < 0.05 threshold of significance
Statistical Analysis 2: Comparison: Control Group; Pretreatment (Baseline) compared to post-treatment (follow-up) CD3 cell density; Test type: Superiority or Other; p = 0.46, t-test, 2 sided — P < 0.05 threshold of significance
Statistical Analysis 3: Comparison: Rituximab Group; pretreatment (baseline) compared to post-treatment (follow-up) biopsy CD20 cell density; Test type: Superiority or Other; p = 0.054, t-test, 2 sided — P < 0.05 threshold of significance
Statistical Analysis 4: Comparison: Control Group; Pretreatment (baseline) compared to post-treatment (follow-up) CD20 cell density; Test type: Superiority or Other; p = 0.62, t-test, 2 sided — P < 0.05 threshold of significance

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Rituximab Group: Rituximab Group: Rituximab infusion day 1 and day 14.
- Control Group: No Rituximab; Standard maintenance immunosuppressive regimen only.
Arm/Group | Rituximab Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

LIMITATIONS AND CAVEATS:
The limitations were small number of participants and short follow up time of only 12 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No